CLINICAL TRIAL: NCT05309538
Title: Effect of Modified Epley's & Semont's Maneuvers With or Without Beta-histine on Benign Paroxysmal Positional Vertigo: A Randomized Control Trail
Brief Title: Paroxysmal Positional Vertigo & Repositioning Maneuvers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 336
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: BPPV
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo | interventions — Betahistine

STUDY DESIGN:
Intervention Model Description: 2 groups , group A contro group and group B experimental group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Control group
  Interventions: Other: Modified eply & Semont maneuver
- group B (Experimental): experimental group
  Interventions: Other: betahistine & Modified eply & Semont maneuver

INTERVENTIONS:
Other: Modified eply & Semont maneuver — repositioning maneauvers
  Arms: Group A
Other: betahistine & Modified eply & Semont maneuver — antihistamine plus repositioning maneuvers
  Other Names: Modified eply & Semont maneuver
  Arms: group B

SUMMARY:
: Benign Paroxysmal Positional Vertigo is a condition related to vestibular system accompanied by dizziness, tinnitus and balance problems leading to increased fall risk and potential disability. Various treatment options are available including pharmacotherapy and vestibular rehabilitation with varied results

DETAILED DESCRIPTION:
Objective: The objective of this study was to compare the efficacy of Modified Epley & Semont's maneuver with and without Betahistine for BPPV Material & Methods: The study was a single blind randomized control trail. Total number of patients were 97 as calculated by Epitool calculator. Duration of the study was of one year from 2 January 2021 to 1st January 2022. Out of a total 97 patients, 90 met the inclusion criteria. These participants were randomized by lottery method into two equal groups. Group A (control group) was receiving both maneuvers only while group B (experimental group) included participants receiving betahistine along with both maneuvers. The impact of dizziness and quality of life was measured through EQ-5D-5L questionnaire and dizziness handicap inventory (DHI) in order to analyze the effectiveness of treatments. Pre and Post treatment results were compared within group by Wilcoxon rank test and for between groups, Mann Whitney U test was performed

ELIGIBILITY:
Inclusion Criteria:

* age between 18-60
* positive modified Dix Hil pike test
* repetitive vertigo spells affecting activities of daily livings (ADLs)

Exclusion Criteria:

* any cervical spine problem
* vertigo due to central disease
* tumors
* systemic disease
* cardiac disease
* Parkinson disease
* bed bound patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
DHI | 1 month
  dizziness handicap inventery
EQ-5D-5L | 1 month
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD SALMAN, M.Phil*, Principal Investigator — the neurocouncil hospital
Locations (1):
- the Neurocouncil Clinic, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
we would share with other researcher so that they might be able to find study gaps

REFERENCES:
- [Background] You P, Instrum R, Parnes L. Benign paroxysmal positional vertigo. Laryngoscope Investig Otolaryngol. 2018 Dec 14;4(1):116-123. doi: 10.1002/lio2.230. eCollection 2019 Feb. PMID 30828628
- [Background] Kerber KA, Burke JF, Skolarus LE, Meurer WJ, Callaghan BC, Brown DL, Lisabeth LD, McLaughlin TJ, Fendrick AM, Morgenstern LB. Use of BPPV processes in emergency department dizziness presentations: a population-based study. Otolaryngol Head Neck Surg. 2013 Mar;148(3):425-30. doi: 10.1177/0194599812471633. Epub 2012 Dec 21. PMID 23264119
- [Background] Kitanaka J, Kitanaka N, Hall FS, Amatsu Y, Hashimoto K, Hisatomi E, Kitao E, Mimura M, Nakamura M, Ozawa R, Sato M, Tagami K, Uhl GR, Takemura M. In vivo evaluation of effects of histamine H3 receptor antagonists on methamphetamine-induced hyperlocomotion in mice. Brain Res. 2020 Aug 1;1740:146873. doi: 10.1016/j.brainres.2020.146873. Epub 2020 May 5. PMID 32387137